CLINICAL TRIAL: NCT03983863
Title: Mapping Institutional Identities and the Production of Ethics
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999919106; 19-HG-N106
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: IRB Decision Making
Keywords: NIH; Panel; Member/Staff; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IRB: Our target study population consists of all members/staff of NIH IRBs and IRB panels that fall under the NIH Intramural Federal Wide Assurance (FWA).

SUMMARY:
Background:

Researchers want to learn how members of IRB committees interact with each other. They want to see how this affects the decision-making process. They want to learn how members see their role and the roles of their fellow members. They want to see if these views are actualized during meetings. To do this, researchers will sit in on IRB meetings and interview committee members.

Objective:

To explore the dynamics between IRB members. To explore how these dynamics affect the IRB process of decision making.

Eligibility:

NIH IRB staff or members

Design:

In Phase I, an investigator (AI) will sit in on IRB meetings for 6 months. The AI will take notes on the dynamics of the committees. The AI s will focus will be on the dialogue and the behavior of both the group and each member. The AI will also focus on the factors that form the decision-making process. The AI will audio-record the meetings to help take detailed notes. These recordings will be destroyed after 3 months.

If the AI does not hear from members before the IRB meetings, the AI will assume that the member is agreeing to take part in Phase I.

In Phase II, the AI will contact some members about taking part in a 60-minute interview. The interview will be semi-structured. It will be on site and in person. It will explore how the members see their role and the roles of others on the committee.

Contact information will be collected only for members who take part in Phase II.

Data will be de-identified.

Withdrawing from the study will not affect any member s role on the IRB.

DETAILED DESCRIPTION:
Objective: The study has two objectives. The primary objective is to explore what dynamics exist within IRB committees, how members in each role interact with each other, and how these interactions affect participation in the deliberation/decision-making process.

The secondary objective of this research is to explore what each member/staff perceives his/her role and the roles of other committee members to be and whether these perceptions are congruent with how roles are actualized during meetings.

Study Population: Our target population consists of all members/staff of NIH IRBs and IRB panels that fall under the NIH Intramural Federal Wide Assurance (FWA).

Design: The project will involve two phases: direct observation and semi-structured interviews. Phase I (direct-observations) will involve an associate investigator, Hina Walajahi, sitting in on regularly scheduled IRB meetings at the NIH and taking observational notes on committee dialogue, individual and group behavior, and factors that contribute to the decision-making process. Meetings will be audio-recorded in order to validate the observation notes. The observational data will be used to select appropriate committee members/staff and guide questions for the semi-structured interviews.

For Phase II (semi-structured interviews), the same associate investigator will conduct in-person, semi-structured interviews with contacted IRB members/staff regarding role perception respective to other members and the committee as a whole. Interviews will last approximately 60 minutes. They will be audio-recorded and transcribed.

Outcome Measures: A qualitative codebook will be created from observational and interview data, focusing on themes including, but not limited to: member interactions, member participation in discussion, committee deliberation processes and voting behavior.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

All members/staff of NIH IRBs and IRB panels that fall under the NIH Intramural Federal Wide Assurance (FWA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All members/staff of NIH IRBs and IRB panels that fall under the NIH Intramural Federal Wide Assurance (FWA).@@@
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Dynamics | Enrollment
  The primary objective is to explore what dynamics exist within IRB committees, how members in each role interact with each other, and how these interactions affect participation in the deliberation/decision-making process. This will be explored through direct observation of IRB committee meetings.

SECONDARY OUTCOMES:
Perception | Single follow-up session
  The secondary objective of this research is to explore what each member/staff perceives his/her role and the roles of other committee members to be and whether these perceptions are congruent with how roles are actualized during meetings. This will be explored through semi-structured interviews with select IRB committee members/staff.

CONTACTS AND LOCATIONS:
Overall Officials: Sara C Hull, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States